CLINICAL TRIAL: NCT06934889
Title: Phase Ib Trial of ABBV-637 or ABBV-155 in Combination With ERAS-801 for Glioblastoma With Amplification of the Epidermal Growth Factor Receptor
Brief Title: Study of ABBV-637 or ABBV-155 With ERAS-801 for People With Glioblastoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-409
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma; Gliosarcoma
Keywords: WHO grade IV; ABBV-637; ABBV-155; ERAS-801; 24-409
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Temozolomide; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Phase Ib Trial of ABBV-637 or ABBV-155 in Combination with ERAS-801. The first eight patients were randomized 1:1 to: ABBV-637 or ABBV-155 (6 to cohorts A/B and 2 to cohorts C/D) using the Randomization Module in the Clinical Research Database (CRDB). Due to drug viability and impending expiration dates, the trial will no longer use randomization going forward beginning with patient 9. Participants will be assigned.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort A (Recurrent) (Experimental): will receive ABBV-637 before standard surgery, followed by ABBV-637 and ERAS-801 after standard surgery.
  Interventions: Drug: ERAS-801; Drug: ABBV-637
- Cohort B (Recurrent) (Experimental): will receive ABBV-155 before standard surgery, followed by ABBV-155 and ERAS-801 after standard surgery
  Interventions: Drug: ERAS-801; Drug: ABBV-155
- Cohort C (Newly Diagnosed) (Experimental): will receive ABBV-637 in combination with standard radiation and chemotherapy drug temozolomide.
  Interventions: Drug: ABBV-637; Drug: Temozolomide; Radiation: Radiotherapy
- Cohort D (Newly Diagnosed) (Experimental): will receive ABBV-155 in combination with standard radiation and chemotherapy drug temozolomide
  Interventions: Drug: ABBV-155; Drug: Temozolomide; Radiation: Radiotherapy

INTERVENTIONS:
Drug: ERAS-801 — will be administered orally at the assigned dose once daily starting on Cycle 1 Day 1.
  Arms: Cohort A (Recurrent); Cohort B (Recurrent)
Drug: ABBV-637 — will be administered intravenously over one hour (+/- 10 min) once every 28 days on the first day of the new cycle.
  Arms: Cohort A (Recurrent); Cohort C (Newly Diagnosed)
Drug: ABBV-155 — will be administered intravenously over at least 30 minutes once every 21 days on the first day of the new cycle.
  Arms: Cohort B (Recurrent); Cohort D (Newly Diagnosed)
Drug: Temozolomide — Temozolomide will be continued for 6 cycles after radiation.
  Arms: Cohort C (Newly Diagnosed); Cohort D (Newly Diagnosed)
Radiation: Radiotherapy — will be given as per standard of care radiation for GBM
  Arms: Cohort C (Newly Diagnosed); Cohort D (Newly Diagnosed)

SUMMARY:
The researchers are doing this study to find out whether the drugs ABBV-637 and ABBV-155 are safe treatments that cause few or mild side effects when given alone or in combination with ERAS-801 in people with recurrent GBM.

DETAILED DESCRIPTION:
Stage 1 will run first, during which patients will be randomized to either Cohort A or B if recurrent GBM, and Cohort C or D if newly diagnosed. After these 4 cohorts are complete, and if the combinations have been safe and tolerable, the combination will be further evaluated in Stage 2.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older at the time of consent signing.
* All Patients must have WHO Grade IV Glioblastoma/Gliosarcoma using WHO 2021 criteria and include the diagnosis of molecular GBM, recurrent patients must be progressive or recurrent following radiation therapy +/- chemotherapy
* Patients must be IDH wild type by CLIA-certified laboratory assay available at time of consent.
* Patients must have evidence of EGFR gene amplification by CLIA-certified laboratory assay at time of consent.
* Patients must have measurable disease as per RANO criteria pre-operatively (there is no requirement for post-operative disease to be present or absent). [cohort A/B only]
* Patients must be able to tolerate MRIs
* Patients may have no more than 2 prior therapy regimens. [cohort A/B only]
* Patients must have recovered from severe toxicity of prior therapy. The following intervals from previous treatments are required to be eligible:

  1. 12 weeks from the completion of radiation
  2. 6 weeks from a nitrosourea chemotherapy
  3. 3 weeks from a non-nitrosourea chemotherapy
  4. 4 weeks from any investigational (not FDA-approved) agents
  5. 6 months from the last treatment with bevacizumab
  6. 2 weeks or 5 half-lives from administration of a non-cytotoxic, Chemotherapies other than bevacizumab, whichever is shorter
* Patients must be undergoing surgery that is clinically indicated as determined by their care providers. [cohort A/B only] Patients must be eligible for surgical resection according to the following criteria:

  a. Expectation that the surgeon is able to resect at least 500 mg of tumor from enhancing tumor with low risk of inducing neurological injury.
* Paraffin embedded tissue must be available from initial surgical resection at diagnosis (prior to any treatment). The following amount of tissue is requested: 1 formalin-fixed, paraffin embedded (FFPE) tissue block (preferred) or 10 FFPE unstained slides (5µm thick).
* Patients must have a Karnofsky Performance Status (KPS) ≥60% (i.e. the patient must be able to care for himself/herself with occasional help from others).
* Patients must have the following organ and marrow function:

  1. Absolute neutrophil count >1,200/mcL
  2. Platelets >100,000/mcL
  3. Hemoglobin > 9 g/dL .
  4. Total bilirubin ≤ institutional upper limit of normal, or ≤ 3.0 mg/dL for subjects with Gilbert's syndrome
  5. AST (SGOT) and ALT (SGPT) ≤ 3 × institutional upper limit of normal
  6. Creatinine ≤ institutional upper limit of normal OR Creatinine clearance >60 ml/min/1.73m2 for patients with creatinine levels above institutional normal
  7. APTT/PTT ≤ 1.5 x institutional upper limit of normal
* Echocardiogram with ejection fraction ≥ 50% and no other clinically significant finding that, in the opinion of the investigator, would increase the subject's susceptibility to cardiac toxicity.

  a. If ECHO cannot be performed for structural or safety reasons, a MUGA may be obtained instead after discussion with treating investigator.
* Patients must have a 12-lead electrocardiogram performed within 2 weeks of treatment start with QT interval corrected for heart rate (QTc) < 450 msec (using Fridericia's correction), and no clinically significant abnormalities. (Cohorts A, B, E & F only)
* Women of childbearing potential must have a negative serum pregnancy test prior to study entry. Women of childbearing potential and men treated or enrolled on this protocol must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 4 months after completion of treatment administration. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* A negative serum pregnancy test for all female subjects (except postmenopausal) at the screening visit and a negative urine pregnancy test for all female subjects (except postmenopausal) at baseline before the first dose of study drug.
* If female, subject must be either postmenopausal, OR permanently surgically sterile OR, for women of childbearing potential, practicing at least 1 protocol-specified method of birth control that is effective from study Day 1 through at least 4 months after the last dose of study drug.
* If male, and subject is sexually active with female partner(s) of childbearing potential, he must agree from study Day 1 through 4 months after the last dose of study drug to practice the protocol-specified contraception.
* If female, subject must not be pregnant, breastfeeding, or considering becoming pregnant during the study while receiving study drug and for at least 4 months after the last dose of study drug.
* If male, subject must not be considering fathering a child or donating sperm during the study or for 4 months after the last dose of study drug.
* No known active viral hepatitis infection (including hepatitis B and C) or human immunodeficiency virus (HIV) with the following exceptions:

  * Subjects with a history of hepatitis B that is considered cured may be enrolled at the discretion of the treating investigator.
  * Subjects with a history of hepatitis C that is considered cured with definitive therapy may be enrolled at the discretion of the treating investigator.
  * Subjects with HIV and undetectable viral load, so long as ongoing antiretroviral therapy does not pose risk of adverse drug-drug interactions, at the discretion of the treating investigator.
* Patients must have no concurrent malignancy that requires active therapy.
* Patients must be able to swallow medication by mouth, either tablets or dispersed in solution.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to any of the investigational agents are ineligible.
* Patients with prior therapy with EGFR targeting agents are ineligible because treatment with EGFR kinase inhibitors or other EGFR-targeted agents has the potential to deplete the tumor of EGFR-amplified or EGFR mutant cell populations and confound the evaluation of the investigational regimen. Patients would only be eligible if surgery on a recurrence after the EGFR-targeted therapy confirmed persistence of an EGFR alteration.
* Patients on enzyme-inducing anti-epileptic drugs (EIAED) are not eligible for treatment on this protocol. Patients may be on non-enzyme inducing anti-epileptic drugs or not be taking any anti-epileptic drugs. Patients previously treated with EIAED may be enrolled if they have been off the EIAED for 10 days or more prior to the first dose of study drug(s).
* Patients must not have evidence of significant hematologic, renal, or hepatic dysfunctioPatients must not have evidence of significant intracranial hemorrhage (For example, in the recurrent setting, circumstances where the intracranial hemorrhage would obscure the amount and quality of tissue obtained at the time of the on-treatment surgery).
* Patients with uncontrolled intercurrent illness including, but not limited to, hypertension, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/ social situations that would limit compliance with study requirements, are ineligible.
* Participants with clinically significant cardiovascular disease including, but not limited to:

  * No recent history (within 6 months) of congestive heart failure (defined as New York Heart Association, Class 2 or higher), ischemic cardiovascular event, cardiac arrhythmia requiring pharmacological or surgical intervention, pericardial effusion, or pericarditis.
  * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG, e.g., complete left bundle branch block, second- or third-degree heart block, PR-interval > 250 ms.
  * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, or any concomitant medication know to prolong the QT interval.
* No history of clinically significant medical and/or psychiatric conditions or any other reason that, in the opinion of the investigator, would interfere with the subject's participation in this study or would make the subject an unsuitable candidate to receive study drug
* Pregnant women are excluded from this study because the investigational regimens have potential for teratogenic or abortifacients effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated on this study.
* HIV-positive patients on strong CYP3A4 inducers or inhibitors are ineligible because of the potential for pharmacokinetic interactions.
* Patients who have acute or currently active/requiring anti-viral therapy hepatic or biliary disease are ineligible (with the exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases from the primary brain tumor, or stable chronic liver disease per investigator assessment).
* Patients receiving P-gp inhibitors/P-gp substrates with narrow therapeutic index are ineligible.
* Patients who are receiving a drug that has a risk of QTc prolongation with known risk of if QTc is ≥ 460 msec. are ineligible. (Temozolomide is allowed for cohorts C,D, E and F)
* Subject must not have systemically used known moderate or strong cytochrome P450 (CYP)3A inhibitors within 10 days before the first dose of study drug and throughout the study.
* Subject must not have received any live vaccine within 2 weeks before the first dose of study drug, or be expected to need a live vaccination during study participation including at least 4 weeks after the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 1 year
  All patients who receive a single dose of investigational drug will be included in the primary endpoint analysis. Will be measured descriptively using CTCAE v5.0

SECONDARY OUTCOMES:
Overall survival | 1 year
  Overall survival will be defined from pre-surgical treatment start date to date of death due to any cause.
Progression-free survival (PFS) | 6 months
  Progression-free survival will be defined from pre-surgical treatment start date to date of progression or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kaley, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - University of Miami (Data collection only), Miami, Florida
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm